CLINICAL TRIAL: NCT05846087
Title: Mobile App-delivered Sleep Therapy (SleepFix) for Individuals With Chronic Low Back Pain and Insomnia: a Randomized Controlled Trial With Internal Pilot Study
Brief Title: Mobile App-delivered Sleep Therapy (SleepFix) for Individuals With Chronic Low Back Pain and Insomnia
Acronym: SleepBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: Cooperative Research Centre for Alertness, Safety and Productivity (Unknown); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X23-0145
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low-back Pain; Insomnia
Keywords: low back pain; insomnia; digital behavioral therapy for insomnia; sleep retraining therapy; pain interference
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Low Back Pain

STUDY DESIGN:
Intervention Model Description: open labelled, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Researchers responsible for randomization and data-analysis will be blinded to the study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Three weeks of sleep retraining therapy - behavioral component of cognitive behavioral therapy for insomnia. This will be self-delivered by participants digitally using the smart phone App 'SleepFix'.
  Interventions: Behavioral: sleep retraining therapy
- Control (Active Comparator): Sleep health education modules delivered each week for three weeks. Modules contain information about sleep and insomnia; how insomnia affects other aspects of life; what activities influence health sleep (sleep hygiene) and information designed to dispel false beliefs about sleep
  Interventions: Other: sleep health education modules

INTERVENTIONS:
Behavioral: sleep retraining therapy — Sleep retraining therapy improves sleep efficiency (total sleep time/total time in bed) by reducing the amount of time spent in bed awake. The digitally designed version which SleepFix delivers uses an algorithm which requires the users current sleep times and ideal wake-up time to determine when one should get into bed to fall asleep and when one should get out of bed.
  Other Names: sleep restriction therapy; sleep consolidation therapy
  Arms: Treatment
Other: sleep health education modules — educational modules about sleep and insomnia; its causes; and its impact on various aspects of life. This information is arranged into three modules which will be provided to participants over three weeks.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the efficacy of a digital behavioral therapy for insomnia (dBTi) in people with chronic low back pain and insomnia. The main question it aims to answer is whether a 3 week period of dBTi can improve pain-related interference 6 weeks from commencement.

Researchers will compare the treatment (dBTi) to an active control (Sleep health education modules) to see if there is a significant difference in outcomes at baseline and end-of-study (6 weeks).

DETAILED DESCRIPTION:
This study is an online, open-labelled, two-arm, parallel-group randomized controlled trial with embedded internal pilot study of dBTi (SleepFix) versus sleep health education control in adults with chronic low back pain (LBP) and insomnia.

To be enrolled in the study, participants are required to complete online pre-screening survey followed by a telephone screening interview with further questions and to verbally explain to participants what is required of them in this study. After interview screening, participants will receive an online baseline questionnaire to complete. Once completed, participants will be randomised to one of two study arms. The treatment arm consists of a dBTi intervention using the SleepFix mobile application. The dBTi intervention takes a minimum of 3 weeks to complete with participants allowed to use SleepFix for longer if they wish. Participants randomized to the control arm will be provide sleep health education through email released weekly during the 3-weeks of intervention treatment. Treatment control participants will receive access to SleepFix once end-of-study questionnaire has been completed.

The study will be conducted online via secure platforms with recruitment primarily through social media advertisements. The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Glebe, NSW, 2037, Australia.

Phase 1 of the study is an internal pilot study which will assess the feasibility of recruitment, data collection and reporting. The following stop-go progression criteria will be used to determine whether we proceed to phase 2 which will continue recruitment until the sample size is reached (n = 134) to determine our primary outcomes. We will:

1. Go if >40% of total sample size (n = 54) are randomized to study arms within 6-months from recruitment start date.
2. Stop if >40% of randomized participants fail to complete week 6 end-of-study questionnaires at 6 months from recruitment start date.

Participants who complete the treatment arm of the study will be invited to take part in a post-study interview exploring the user experience of SleepFix and whether it has led to any changes in pain and sleep management. We are conducting these interviews to understand qualitatively how this population feels towards SleepFix and their feelings towards the importance of sleep for their chronic LBP condition.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years.
2. Chronic low back pain (pain in lower back region which has been present for 3 months or more).
3. Able to give informed online consent.
4. Insomnia Severity Index Score >10.
5. English fluency.
6. Access to a smartphone and willingness/proficiency to use a mobile app for healthcare.

Exclusion Criteria:

1. Currently experiencing sciatica or other neuropathic pain condition OR inflammatory condition of the spine/vertebral column.
2. Shift-workers. Regular work that falls outside the hours between 7am and 6pm.
3. Trans-meridian travel to a destination with >2 hours' time-difference (within last 7-days and will subjective reports that they are not experiencing jet lag).
4. Serious medical and/or psychiatric illnesses/disorders (e.g. Major Depressive Disorder, epilepsy, bipolar disorder, heart failure, dementia).
5. Sleep disorders (includes: Obstructive Sleep Apnoea, Sleep Behaviour Disorder (i.e sleep talking/walking, REM), Circadian Rhythm Disorder, Restless leg syndrome, Narcolepsy or Bruxism).
6. Sleep devices (e.g. CPAP)
7. Currently receiving psychotherapy for insomnia including Cognitive Behavioural Therapy (CBT).
8. Professional driver or operate heavy machinery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Female
  2. Male
  3. Non-binary
  4. Prefer not to say
Enrollment: 106 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Pain interference | 6 weeks
  Brief Pain Inventory (BPI) - pain interference is a subscale of the BPI consisting of 7 items which assess the extent to which pain interferes with: general activity; mood; walking; work (at home or outside); relationships; sleep; and enjoyment of life. BPI items are reported using an 11-point Likert type scale. (0 = "does not interfere"; 10 = "interferes completely"). Responses are summed to provide a global interference score between 0 and 70.

SECONDARY OUTCOMES:
Pain intensity | 6 weeks
  Brief Pain Inventory (BPI) - pain intensity is a subscale of the BPI which is composed of 4-items which ask a rating for current pain, average pain, worst and least pain over the past 24 hours using an 11-point Likert type scales (0 = "No pain at all"; 10 = "worst pain possible").
Insomnia severity index (ISI) | 6 weeks
  7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 4) regarding symptoms over the past 2 weeks. All items are summed with total scores ranging from 0-28.
Pittsburgh Sleep Quality Index (PSQI) | 6 weeks
  19-item self-reported questionnaire which, in this case, assesses sleep quality and disturbances over the previous 2 weeks so only variables across a time-period not including the therapy window are measured. Seven component scores are derived from the responses, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0-21) where a score of 5 or more indicates poor sleep quality.
Pain-related beliefs and attitudes about sleep (PBAS) | 6 weeks
  The pain-related beliefs and attitudes about sleep questionnaire (PBAS) is a 10-item self-reported measure developed for assessment and treatment of insomnia comorbid with chronic pain. PBAS assesses one's beliefs about the interaction of pain and sleep. Items are measured on an 11-point likert type scale (0 = "strongly disagree"; 10 = "strongly agree").
Patient Health Questionnaire-2 (PHQ-2) | 6 weeks
  The Patient Health Questionnaire-2 is a 2-item self-reported measure of depressive symptoms over the past 2 weeks. Participants are asked to answer questions about the severity of depressive symptoms. Scores for each question (Likert type scale "not at all" = 0 to "nearly every day" = 3) sum to a total score of 0 to 6.
General Anxiety Disorder-7 (GAD-7) | 6 weeks
  The General Anxiety Disorder-7 (GAD-7) is a 7-item self-administered scale used to assess the severity of generalised anxiety by asking how often participants have experienced symptoms in the previous two weeks. It consists of a three-point Likert type scale for each item (ranging from "not at all" = 0 to "nearly every day" = 3). All items are summed with total scores ranging from 0-21 where 5, 10 and 15 indicate the cut-off scores for mild, moderate and severe anxiety, respectively.
EuroQol five-dimensional (EQ-5D) | 6 weeks
  The EuroQol five-dimensional (EQ-5D) is a well-validated, generic instrument for measuring health related quality of life at the time of completion. The self-reported questionnaire is comprised of 2 components including: (1) Health state description - measured in terms of 5 dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression and (2) evaluation - where participants are asked to evaluate their overall health using a visual analogue scale. In Part 1, each item is assigned a level (ranging from "indicating no problem"1 - "indicating unable to/extreme problems" - 5) according to the response and this descriptive data is used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gordon, A/Prof, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
The trial investigators will be given access to the cleaned data set. The project data set will be housed online in the study web portal created for the study, and all data will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.
  Data will not be shared without permission of Principal Investigators. All data available for sharing will be stored on a web-based database located in Australia. After the study, a non-identified dataset may be made available online in a data repository.

REFERENCES:
- [Background] Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Transl Med. 2020 Mar;8(6):299. doi: 10.21037/atm.2020.02.175. PMID 32355743
- [Background] Kelly GA, Blake C, Power CK, O'keeffe D, Fullen BM. The association between chronic low back pain and sleep: a systematic review. Clin J Pain. 2011 Feb;27(2):169-81. doi: 10.1097/AJP.0b013e3181f3bdd5. PMID 20842008
- [Background] Bilterys T, Siffain C, De Maeyer I, Van Looveren E, Mairesse O, Nijs J, Meeus M, Ickmans K, Cagnie B, Goubert D, Danneels L, Moens M, Malfliet A. Associates of Insomnia in People with Chronic Spinal Pain: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Jul 19;10(14):3175. doi: 10.3390/jcm10143175. PMID 34300341
- [Background] Amiri S, Behnezhad S. Sleep disturbances and back pain : Systematic review and meta-analysis. Neuropsychiatr. 2020 Jun;34(2):74-84. doi: 10.1007/s40211-020-00339-9. Epub 2020 Mar 12. PMID 32166629
- [Background] Cheatle MD, Foster S, Pinkett A, Lesneski M, Qu D, Dhingra L. Assessing and Managing Sleep Disturbance in Patients with Chronic Pain. Sleep Med Clin. 2016 Dec;11(4):531-541. doi: 10.1016/j.jsmc.2016.08.004. Epub 2016 Oct 27. PMID 28118876
- [Background] Aji M, Glozier N, Bartlett D, Peters D, Calvo RA, Zheng Y, Grunstein R, Gordon C. A feasibility study of a mobile app to treat insomnia. Transl Behav Med. 2021 Mar 16;11(2):604-612. doi: 10.1093/tbm/ibaa019. PMID 32227087
- [Background] Irish LA, Kline CE, Gunn HE, Buysse DJ, Hall MH. The role of sleep hygiene in promoting public health: A review of empirical evidence. Sleep Med Rev. 2015 Aug;22:23-36. doi: 10.1016/j.smrv.2014.10.001. Epub 2014 Oct 16. PMID 25454674
- [Background] Howarth A, Quesada J, Silva J, Judycki S, Mills PR. The impact of digital health interventions on health-related outcomes in the workplace: A systematic review. Digit Health. 2018 May 10;4:2055207618770861. doi: 10.1177/2055207618770861. eCollection 2018 Jan-Dec. PMID 29942631
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Aji M, Gordon C, Stratton E, Calvo RA, Bartlett D, Grunstein R, Glozier N. Framework for the Design Engineering and Clinical Implementation and Evaluation of mHealth Apps for Sleep Disturbance: Systematic Review. J Med Internet Res. 2021 Feb 17;23(2):e24607. doi: 10.2196/24607. PMID 33595441
- [Background] Mameli S, Pisanu GM, Sardo S, Marchi A, Pili A, Carboni M, Minerba L, Trincas G, Carta MG, Melis MR, Agabio R. Oxytocin nasal spray in fibromyalgic patients. Rheumatol Int. 2014 Aug;34(8):1047-52. doi: 10.1007/s00296-014-2953-y. Epub 2014 Feb 8. PMID 24509894
- [Background] Tang NK, Goodchild CE, Sanborn AN, Howard J, Salkovskis PM. Deciphering the temporal link between pain and sleep in a heterogeneous chronic pain patient sample: a multilevel daily process study. Sleep. 2012 May 1;35(5):675-87A. doi: 10.5665/sleep.1830. PMID 22547894
- [Background] Roth SH, Fleischmann RM, Burch FX, Dietz F, Bockow B, Rapoport RJ, Rutstein J, Lacouture PG. Around-the-clock, controlled-release oxycodone therapy for osteoarthritis-related pain: placebo-controlled trial and long-term evaluation. Arch Intern Med. 2000 Mar 27;160(6):853-60. doi: 10.1001/archinte.160.6.853. PMID 10737286
- [Background] Malfliet A, Bilterys T, Van Looveren E, Meeus M, Danneels L, Ickmans K, Cagnie B, Mairesse O, Neu D, Moens M, Goubert D, Kamper SJ, Nijs J. The added value of cognitive behavioral therapy for insomnia to current best evidence physical therapy for chronic spinal pain: protocol of a randomized controlled clinical trial. Braz J Phys Ther. 2019 Jan-Feb;23(1):62-70. doi: 10.1016/j.bjpt.2018.10.007. Epub 2018 Oct 29. PMID 30389347
- [Background] Kean J, Monahan PO, Kroenke K, Wu J, Yu Z, Stump TE, Krebs EE. Comparative Responsiveness of the PROMIS Pain Interference Short Forms, Brief Pain Inventory, PEG, and SF-36 Bodily Pain Subscale. Med Care. 2016 Apr;54(4):414-21. doi: 10.1097/MLR.0000000000000497. PMID 26807536
- [Background] Jungquist CR, O'Brien C, Matteson-Rusby S, Smith MT, Pigeon WR, Xia Y, Lu N, Perlis ML. The efficacy of cognitive-behavioral therapy for insomnia in patients with chronic pain. Sleep Med. 2010 Mar;11(3):302-9. doi: 10.1016/j.sleep.2009.05.018. Epub 2010 Feb 4. PMID 20133188
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Afolalu EF, Moore C, Ramlee F, Goodchild CE, Tang NK. Development of the Pain-Related Beliefs and Attitudes about Sleep (PBAS) Scale for the Assessment and Treatment of Insomnia Comorbid with Chronic Pain. J Clin Sleep Med. 2016 Sep 15;12(9):1269-77. doi: 10.5664/jcsm.6130. PMID 27448428
- [Background] Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item questionnaire (PHQ-2). J Psychosom Res. 2005 Feb;58(2):163-71. doi: 10.1016/j.jpsychores.2004.09.006. PMID 15820844
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046